CLINICAL TRIAL: NCT00823290
Title: A Phase I Trial of Sorafenib and LBH589 in the Treatment of Advanced HCC
Brief Title: Sorafenib and LBH589 in Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left site
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: PD Dr. Matthias Ocker, University Hospital Erlangen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BDE02
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; sorafenib; HDAC; LBH589; Panobinostat
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sorafenib + LBH589 — Sorafenib standard regimen + oral LBH589

SUMMARY:
Histone deacetylase inhibitors (HDACi) like LBH589 have recently been established as novel potent anti-cancer agents for solid and hematologic malignancies. Several pre-clinical reports have shown a good anti-tumoral activity of different HDACi on human or murine HCC models. These compounds, e.g. Trichostatin A, SAHA, MS-275 and others, have been shown to induce apoptosis in HCC cells and to inhibit growth of HCC by inhibiting proliferation and tumor-related angiogenesis in vivo. Furthermore, HDACi sensitize HCC in a synergistic manner to other forms of cytotoxic stimulation, e.g. by conventional chemotherapeutic drugs or TRAIL-mediated apoptosis. It has also been shown that the combination of HDACi with various kinase inhibitors like sorafenib, erlotinib or others, promotes the anti-tumor efficacy of single agents.

Based on the investigators' own previous experiences with different HDACi and LBH589 in preclinical HCC models, a strong anti-proliferative and pro-apoptotic as well as an anti-angiogenic effect will be expected by combining LBH589 with an existing sorafenib treatment. It is assumed that this combination will prolong overall survival and time-to-progression with lowered adverse effects in HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients > 18 years of age
* patients who have a life expectancy of at least 12 weeks
* patients with advanced hepatocellular carcinoma
* patients with have histologically or radiologically confirmed HCC; documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable
* at least one tumor lesion that can be accurately measured in at least one dimension according to RECIST and which has not been treated with local therapy (hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection); the scans should be approximately 2 weeks old to be used as baseline scan
* patients who received Sorafenib 2 x 400 mg a day between 4 to 6 weeks without dose reduction due to dose limiting toxicities
* at least a period of 4 weeks prior to baseline scan after completion of a local therapy such as surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation
* patients who have an ECOG PS of 0, 1 or 2 respectively Karnofsky Performance Status > 70%
* cirrhotic status of Child-Pugh-class A or B (max. 7 points); Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period
* no signs of decompensated liver cirrhosis
* white blood cells > 3,000/mm³
* neutrophils > 1,500/mm³
* platelets > 100,000/mm³
* bilirubin > 3x upper limit of normal (ULN)
* AST and ALT > 3x ULN
* creatinine normal
* PTT < 1.5x ULN
* fasting serum cholesterol < 350 mg/dL
* triglycerides < 300 mg/dL
* proteinuria < 1g in 24 h
* no history of allergic reactions to compounds similar to Panobinostat or Sorafenib
* no prior thromboembolic disease
* no history of hematemesis or hemoptysis
* no other uncontrolled illness
* women of childbearing potential must have had a negative serum or urine pregnancy test 48 hours prior to the administration of the first study treatment
* patients who give a written informed consent obtained according to local guidelines
* no other concurrent investigational drugs or anticancer agents
* no concurrent traditional Chinese or herbal medicine (e.g. sho-saiko-to, silymarine)

Exclusion Criteria:

* patients currently receiving chemotherapy, immunotherapy or radio-therapy or who have received these within 4 weeks of study entry
* patients who do not tolerate therapy with Sorafenib 2 x 400 mg a day
* prior use of systemic investigational agents for HCC
* previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors and any cancer curatively treated > 3 years prior to entry is permitted;
* chronic treatment with steroids or another immunosuppressive agent
* a known history of HIV seropositivity
* renal failure requiring hemo- or peritoneal dialysis
* history of cardiac disease: congestive heart failure (> New York Heart Association class 2), active coronary artery disease, cardiac arrhythmias requiring anti- arrhythmic therapy other than beta blockers or digoxin, uncontrolled hypertension; myocardial infarction more than 6 month prior to study entry is permitted
* active clinically serious infections (> grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events - CTCAE - version 3.0)
* known carcinomatous meningitis or uncontrolled brain disease
* patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry or on oral anti-vitamin K medication (except low dose coumarin)
* history of organ allograft
* uncontrolled diabetes
* impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption LBH589 or Sorafenib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* patients who have not recovered from surgery
* female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; if barrier contraceptives are being used, these must be continued throughout the trial by both sexes
* patients who are using other investigational agents or who had received investigational drugs > 4 weeks prior to study inclusion
* history of noncompliance to medical regimens
* patients unwilling to or unable to comply with the protocol
* substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of LBH589 | 1 year

SECONDARY OUTCOMES:
Safety, tolerability and adverse events (based on CTCAE 3.0) | 1 year
Reduction of lesion size (radiologically assessed according to RECIST) | 1 year
Laboratory abnormalities (CTC grade 3 or grade 4 toxicities) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, University Hospital Erlangen, Erlangen, Germany